CLINICAL TRIAL: NCT03603886
Title: Telemedicine Pain Control Program for Teens Undergoing Treatment for Cancer
Brief Title: Adolescent Cancer Telemedicine for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Rally Foundation for Childhood Cancer Research (Other); Bear Necessities Pediatric Cancer Foundation (Unknown)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-000223
Record Dates: First submitted 2018-07-11; First posted 2018-07-27 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Waitlist control group receives intervention following waitlist period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Pain Management (Experimental)
  Interventions: Behavioral: Telemedicine Pain Management Intervention (immediate group)
- Waitlist Control (Other): Treatment as usual comparator
  Interventions: Behavioral: Telemedicine Pain Management Intervention (waitlist group, intervention administered following 4-week waitlist period)

INTERVENTIONS:
Behavioral: Telemedicine Pain Management Intervention (immediate group) — Four weekly telemedicine pain management sessions with a trained provider. Intervention will be delivered via video conferencing platform, and each session will last between 30 and 45 minutes. Intervention topics will include: pain psychoeducation, pain coping tools, pain communication, and pain-related stress management.
  Arms: Telemedicine Pain Management
Behavioral: Telemedicine Pain Management Intervention (waitlist group, intervention administered following 4-week waitlist period) — Four week waitlist period during which participants receive treatment as usual. Following the waitlist period, participants will receive the telemedicine pain management intervention:
  Four weekly telemedicine pain management sessions with a trained provider. Intervention will be delivered via video conferencing platform, and each session will last between 30 and 45 minutes. Intervention topics will include: pain psychoeducation, pain coping tools, pain communication, and pain-related stress management.
  Arms: Waitlist Control

SUMMARY:
Pain in adolescents undergoing treatment for cancer is a common problem, often related to treatment or to the cancer itself. Due to increasing outpatient-based cancer treatment, the burden of care and pain management has shifted to the home environment. Yet, there are limited interventions that target the management of pain at home. Adolescence is marked by increased need for independence and social integration, both of which can be impaired by pain or fear of pain. To address unique needs during this developmental period, this study will test a telemedicine program to enhance pain knowledge and pain control strategies in adolescents ages 12-21 years who are undergoing treatment for cancer.

Fifty-six teens will be randomized to an intervention or wait-list control condition. Patients randomized to the waitlist control condition will receive the intervention following completion of the waitlist condition. The intervention will consist of four weekly 30-45 minute telemedicine (online via videoconferencing platform) sessions with a trained social work or psychology provider. Sessions will focus on pain psychoeducation, coping tools, communication, and stress management. Participants will complete online questionnaires assessing pain coping, pain management, and pain-related impairment at pre-intervention, post-intervention, and 1- and 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-21 years
2. At least two months post cancer diagnosis
3. Experienced pain in the past month as defined by at least one pain experience rated >3 on a 0-10 Numeric Rating Scale
4. Access to the internet for intervention sessions
5. Fluent in English (Given that the intervention will be delivered in English, all adolescents will need to be fluent in English to participate.)

Exclusion Criteria:

1. Significant cognitive impairment that may affect their ability to participate

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Attrition rate | Within 7 days of withdrawing from or completing the intervention
  Determined by the percentage of participants who drop out of the study. An attrition rate of 20% or less will indicate feasibility.
Session attendance | Within 7 days of withdrawing from or completing the intervention
  Determined by the number of sessions that participants attend (out of 4 total sessions). To be considered feasible, 80% of participants must have completed at least 3 of the sessions within a 6-week period.
Acceptance (measured via 3 categorical multiple choice questions assessing acceptability, impressions, and helpfulness of intervention) | Within 7 days of completing the intervention
  Intervention will be deemed acceptable if at least 80% of participants rate each question an average of at least "4" ("Agree") on a 5-point scale anchored by "Strongly Disagree" and "Strongly Agree."

SECONDARY OUTCOMES:
Change in pain coping behaviors as assessed by the Pain Coping Questionnaire (PCQ) | At study enrollment (pre-intervention) and between 4 and 6 weeks later (post-intervention for immediate group, post-waitlist period for waitlist group)
  Assessed by the change in the total score on the 'Coping with Pain' section of the Pain Coping Questionnaire (PCQ) from pre-intervention to post-intervention (immediate group) or post-waitlist period (waitlist group). Calculated by subtracting the pre-intervention score from the post-intervention score. The 'Coping with Pain' section of the PCQ consists of 39 items. The total score is calculated as a mean rating and can range from 1-5 and higher scores indicate greater use of coping strategies.
Change in pain-related impairment as assessed by the PROMIS Pain Interference - Pediatric Short Form v2.0 | At study enrollment (pre-intervention) and between 4 and 6 weeks later (post-intervention for immediate group, post-waitlist period for waitlist group)
  Assessed by the change in the total score on the PROMIS Pain Interference - Pediatric Short Form v2.0 from pre-intervention to post-intervention (immediate group) or post-waitlist period (waitlist group). Calculated by subtracting the pre-intervention score from the post-intervention score. The PROMIS Pain Interference - Pediatric Short Form v2.0 is an 8-item measure whose total score can range from 8-40. Higher scores indicate higher interference caused by pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie K Zeltzer, MD, Principal Investigator — UCLA Pediatric Pain and Palliative Care Program
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States